CLINICAL TRIAL: NCT06080477
Title: Enhancing Post-acute Mental Health Outcomes for Patients With Psychosis in Malawi Through Nurse-delivered Community-based Rehabilitation: The ENHANCE Pilot Trial
Brief Title: Enhancing Mental Health Outcomes for Patients With Psychosis in Malawi Through Community-based Rehabilitation
Acronym: ENHANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-1665; R34MH131234 (NIH)
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: Two-arm individually randomized trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted ENHANCE Intervention (Experimental): Nurse-delivered community-based treatment model for people living with psychosis in the community, coordinated with the usual outpatient care
  Interventions: Behavioral: Adapted ENHANCE Intervention
- Enhanced usual care (Active Comparator): Continue with usual outpatient care, enhanced with additional feedback and clinical recommendations to the outpatient treatment team
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Enhanced Usual Care — Participants randomized to usual care will continue to receive their standard clinical care at Queen Elizabeth Central Hospital (QECH) as previously. The clinical team will be provided a summary of the results of the eligibility assessment, specifically an interpretation of the scores on the symptomatology and disability scales with any relevant clinical recommendations. These individuals will receive no home-based services.
  Arms: Enhanced usual care
Behavioral: Adapted ENHANCE Intervention — Participants randomized to the intervention arm will receive community-based rehabilitation (CBR) delivered by the Queen Elizabeth Central Hospital (QECH) clinical team of psychiatric nurses. The ENHANCE CBR intervention will consist of nurse-delivered home visits over approximately a 12-month period with decreasing intensity, with approximately weekly visits for an initial phase of 2-4 months; biweekly visits for an intermediate phase of 4-6 months; and monthly for a final transition phase of 3-4 months. The exact schedule and duration of each phase will be individualized by the nurse to the participant based on the participant's initial presentation and their response during the intervention. The intervention team will deliver intervention content with the participant and/or family members and caregivers as appropriate to the module.
  Arms: Adapted ENHANCE Intervention

SUMMARY:
The overall aim of the proposed study is to determine the feasibility, acceptability, fidelity, and preliminary effectiveness of the adapted nurse-led, community-based rehabilitation treatment model for community-dwelling individuals living with psychosis in Blantyre, Malawi using a pilot randomized controlled trial.

DETAILED DESCRIPTION:
Psychosis exacts a heavy morbidity and mortality toll worldwide, but especially in low- and middle-income countries (LMICs). Psychotic disorders are one of the most common presenting complaints for individuals admitted to specialty mental health services in many LMICs. Psychotic disorders typically have onset in early adulthood and a chronic course, meaning patients suffer from many years of poor functionality, disability, and lost productivity. Indeed, psychotic disorders remain among the 15 leading causes of disability globally. The chronicity and severity of psychotic disorders exert a heavy burden on family as relatives frequently have to assume caregiver roles in LMIC where access to formal mental health care is limited.

Despite the significant toll of psychosis in LMICs, treatment options are extremely limited and focus heavily on acute, time-limited inpatient stabilization. This focus fails to consider the demonstrated need for long-term post-acute outpatient treatment and community-based rehabilitation to improve outcomes and prevent relapse. Contextual community factors such as reliable continued access to mental health care, stigma and its negative impact on medication adherence, inadequate support, and family conflict are key risk factors for subsequent relapse upon discharge into the community. Research has recommended the need for community interventions to minimize medication non-adherence and limit relapse and readmission.

Community-based rehabilitation (CBR) directly addresses the need for a concerted approach to post-acute community-based care for people with psychosis in low-resource settings. CBR is a general evidence-based approach for the long-term treatment and support of individuals with a broad range of disabilities in resource-constrained settings that is particularly well suited to address the needs of those with psychosis. CBR aims to improve the quality of life of individuals living with disability by supporting medical care engagement, addressing functional goals, and encouraging social inclusion within their families and communities. CBR is amenable to delivery by a range of personnel and involves collaboration between caregivers, community members, and available public sector services to facilitate the rehabilitation of patients.

Accordingly, in this protocol the investigators will pilot-test an adaptation of the evidence-based Community-Based Rehabilitation (CBR) treatment model specifically to address the needs of community-dwelling individuals with psychosis in Malawi. Specifically, investigators will complete a pilot randomized controlled trial to evaluate the feasibility, acceptability, fidelity, and preliminary effectiveness of the adapted CBR treatment model. This work will provide a critical advance in establishing the evidence base for community-based treatment models for people living with psychosis outside of the context of acute inpatient stabilization so as to enhance rehabilitation, functioning, and quality of life.

ELIGIBILITY:
Inclusion Criteria for PWLE:

* Current outpatient at Queen Elizabeth Central Hospital psychiatry clinic
* Age 18 or older
* Diagnosis of schizophrenia spectrum disorder or clinical presentation of symptoms of hallucinations, delusions or thought disorder that persisted for longer than one month and are accompanied by significant functional impairment
* Resident in Blantyre District
* Not planning to relocate out of Blantyre District in next 12 months
* Has a primary caregiver willing to participate in the study
* Has current elevated symptoms or poor functioning as demonstrated by one or more of:

Positive and Negative Symptoms Scale score ≥58

WHO Disability Assessment Schedule 2.0 score ≥35

Clinical Global Impression Severity score ≥2 (at least mildly ill)

Inclusion Criteria for Caregivers:

* Is a current caregiver for an eligible and consenting patient participant.
* Age 18 or older
* Resident in Blantyre District
* Not planning to relocate out of Blantyre District in next 12 months

Exclusion Criteria for PWLE:

* Not a current outpatient at Queen Elizabeth Central Hospital psychiatry clinic
* Not Age 18 or older
* No diagnosis of schizophrenia spectrum disorder or clinical presentation of symptoms of hallucinations, delusions or thought disorder that persisted for longer than one month and are accompanied by significant functional impairment
* Not a resident in Blantyre District
* Planning to relocate out of Blantyre District in next 12 months
* Does not have a primary caregiver willing to participate in the study
* Does not have current elevated symptoms or poor functioning as demonstrated by one or more of:

Positive and Negative Symptoms Scale score ≥58

WHO Disability Assessment Schedule 2.0 score ≥35

Clinical Global Impression Severity score ≥2 (at least mildly ill)

Exclusion Criteria for Caregivers:

* Is not a current caregiver for an eligible and consenting patient participant.
* Not Age 18 or older
* Not a resident in Blantyre District
* Planning to relocate out of Blantyre District in next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate (Recruitment Feasibility) | Baseline
  This measure is the ability to successfully enroll people with lived experience (PWLE) in the pilot intervention. Feasibility will be evaluated by measuring the recruitment rate (number of patients approached in order to accrue the final sample).
Proportion of participants retained in the study (Retention Feasibility) | 12 months
  Feasibility will be evaluated by measuring the proportion of participants retained in the study (number of patients enrolled at baseline who are still enrolled in the trial through 12 months).
Number of Participants Who Were Either Very Satisfied or Somewhat Satisfied with the Intervention (Intervention Acceptability) | Conclusion of study
  The number of patients who were either very satisfied or somewhat satisfied with the intervention among all participants who received the intervention. Satisfaction will be measured on a 4-point Likert scale where 1 indicates high satisfaction and 4 indicates high dissatisfaction.
Proportion of Completed Intervention Sessions (Intervention Attendance Fidelity) | 12 months
  The total number of intervention sessions completed, out of the number of sessions expected to be completed.

SECONDARY OUTCOMES:
Overall Functioning | 12 months
  Level of functioning will be evaluated using the World Health Organization Disability Assessment Schedule (WHODAS 2.0 12-item version). The WHODAS 2.0 measures general disability related to multiple domains (i.e., understanding and communicating, getting around, self care, getting along with people, life activities, work/school, participation in society). Total scores range from 1 (no disability) to 5 (extreme/cannot do), with higher scores indicating more impairment.
Quality of Life based on Short-Form 8 measure | 12 months
  Quality of life will be evaluated using the Short Form-8 (SF-8). The SF-8 is a shorter, 8-item questionnaire that covers the same eight domains as the full SF-36. The 8 items are scored from 1 (not at all confident) to 5 (very confident). Higher scores are indicative of greater ability to manage symptoms.
Change in psychosis symptoms from baseline | Baseline,12 months
  Change in psychosis symptoms from baseline will be evaluated using the Positive and Negative Symptoms Scale (PANSS). The Positive and Negative Syndrome Scale (PANSS) has three subscales: positive (score range 7-49), negative (score range 7-49), and general psychopathology (score range 16-112). The PANSS positive symptom sub-scale is comprised of 7 items rated on a scale of 1-7, representing positive symptoms of schizophrenia. The PANSS negative symptom subscale is comprised of 7 items rated on a scale of 1-7 representing the negative symptoms of schizophrenia, and the general psychopathology subscale is comprised of 16 items rated on a scale of 1-7 representing symptoms of general psychopathology in mental illness. Scores reported are change in symptoms per week, relative to baseline.
Psychosis Symptom Response | 12 months
  Psychosis symptom response will be defined as a ≥20% reduction in symptoms from baseline as measured using the Positive and Negative Symptoms Scale (PANSS) total score. The Positive and Negative Syndrome Scale (PANSS) has three subscales: positive (score range 7-49), negative (score range 7-49), and general psychopathology (score range 16-112). The PANSS positive symptom sub-scale is comprised of 7 items rated on a scale of 1-7, representing positive symptoms of schizophrenia. The PANSS negative symptom subscale is comprised of 7 items rated on a scale of 1-7 representing the negative symptoms of schizophrenia, and the general psychopathology subscale is comprised of 16 items rated on a scale of 1-7 representing symptoms of general psychopathology in mental illness. Scores reported are change in symptoms per week, relative to baseline.
Psychosis Symptom Remission | 12 months
  Psychosis symptom remission will be defined based on the standard Positive and Negative Symptoms Scale (PANSS) definition of minimal or no symptoms on items G5, G9, N1, N4, N6, and P1-3. The Positive and Negative Syndrome Scale (PANSS) has three subscales: positive (score range 7-49), negative (score range 7-49), and general psychopathology (score range 16-112). The PANSS positive symptom sub-scale is comprised of 7 items rated on a scale of 1-7, representing positive symptoms of schizophrenia. The PANSS negative symptom subscale is comprised of 7 items rated on a scale of 1-7 representing the negative symptoms of schizophrenia, and the general psychopathology subscale is comprised of 16 items rated on a scale of 1-7 representing symptoms of general psychopathology in mental illness. Scores reported are change in symptoms per week, relative to baseline.
Clinical Improvement | 12 months
  Clinical improvement will be evaluated using the Clinical Global Impression-Improvement score (CGI-I). The CGI-I is a 1-7 scale, designed to evaluate improvement through a comparison with the initial assessment of the patient at baseline. Possible ratings range from "very much improved" (score of 1) to "very much worse" (score of 7).
Internalized stigma | 12 months
  Internalized stigma will be evaluated using the Internalized Stigma of Mental Illness Inventory (ISMI). A total score is calculated by taking an average of the responses on the items (range=1 to 4). Higher total scores indicate greater internalized stigma.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Pence, PhD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Queen Elizabeth Central Hosptial, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina at Chapel Hill (UNC).
Time Frame: 9 to 36 months following publication
Access Criteria: The investigator who proposes to use the data has approval from an IRB, IEC, or REB, as applicable, and an executed data use/sharing agreement with UNC.

DOCUMENTS (1):
  • Informed Consent Form (2023-10-17): https://cdn.clinicaltrials.gov/large-docs/77/NCT06080477/ICF_000.pdf